CLINICAL TRIAL: NCT01975805
Title: To Determine the Difference in Positive Bacterial Cultures in Cesarean Sections With 2% Chlorhexidine- Gluconate, 70% Isopropyl Alcohol (Chloraprep) vs. Povidone-iodine 10% (Betadine) Preoperative Surgical Scrub
Brief Title: Chlorhexidine Gluconate Versus Povidone Iodine at Cesarean Delivery: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ramen Chmait, Assistant Professor of Clinical Obstetrics&Gynecology, Pediatrics, and Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTP-09-00380; HS-09-00380 (Other: USC)
Record Dates: First submitted 2013-10-23; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy; Cesarean Section
Keywords: cesarean delivery; chlorhexidine; iodine; skin disinfectant
MeSH Terms: interventions — chlorhexidine gluconate; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine Gluconate (Experimental): Use of Chlorhexidine Gluconate as skin disinfectant for cesarean section.
  Interventions: Other: Chlorhexidine Gluconate
- Povidone Iodine (Experimental): Use of Povidone Iodine as skin disinfectant for cesarean section.
  Interventions: Other: Povidone Iodine

INTERVENTIONS:
Other: Chlorhexidine Gluconate
  Arms: Chlorhexidine Gluconate
Other: Povidone Iodine
  Arms: Povidone Iodine

SUMMARY:
Currently there are no published studies comparing the efficacy of Chloraprep and povidone-iodine in decreasing postoperative- wound infection in cesarean sections. However, there have been studies involving other types of surgery that have compared the efficacy of different types of preoperative cleansing agents in preventing postoperative wound infection. These studies have shown that controversy exists over which antiseptic skin preparation is the most effective for preventing postoperative surgical wound infections. The standard of care at Los Angeles County Hospital for preoperative skin antiseptic in cesarean sections is povidone- iodine 10% (betadine), however many other hospitals have made the transition to using Chloraprep. In an attempt to improve on the current standard of care, we propose a quality improvement prospective randomized study to compare the difference in postoperative wound complications with the use of povidone- iodine and Chloraprep as a preoperative antiseptic in cesarean sections. We hypothesize that Chloraprep will be better than Betadine at reducing the incidence of positive bacterial cultures following cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women greater than 36 weeks gestation presenting for scheduled repeat cesarean sections and scheduled primary cesarean sections
* Ages 18-45
* Written informed consent obtained

Exclusion Criteria:

* Patients who are taking antimicrobial therapy for any reason
* Patient with a known allergy to one or both of the prepping agents
* Patients currently taking immunosuppressant drugs
* Active acute or chronic infection
* Current history of cancer
* Open wounds, skin ulcers, sores, and severe acne
* History of methicillin-resistant staphylococcus aureus colonization or oxacillin-resistant staphylococcus aureus colonization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To compare the difference in the number of positive bacterial cultures at the site of the incision after preoperative cleansing with povidone iodine and Chloraprep. | 3 min-18 days after skin preparation

SECONDARY OUTCOMES:
To compare the difference in postoperative wound infections measured by the presence of purulent drainage, temp greater than 100.4 F, induration at the site of incision with the use of povidone-iodine and Chloraprep. | Post operative days 0-18

CONTACTS AND LOCATIONS:
Overall Officials: Cynelle M. Kunkle, MD, Principal Investigator — University of Southern California; Ramen Chmait, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252